CLINICAL TRIAL: NCT02450799
Title: Corrected VA With Long-Term Follow-Up After AcrySof® IOL Implantation
Brief Title: Corrected VA With Long-Term Follow-Up After AcrySof® Intraocular Lens (IOL) Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: ILQ245-P001; UMIN000017727 (Other: UMIN)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Pseudophakia
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AcrySof IOL (Experimental): Acrylic IOL, prior implantation (1994-2000) in one or both eyes
  Interventions: Device: Acrylic IOL
- Silicone IOL (Active Comparator): Silicone IOL, prior implantation (1994-2000) in one or both eyes
  Interventions: Device: Silicone IOL
- PMMA IOL (Active Comparator): PMMA IOL, prior implantation (1994-2000) in one or both eyes
  Interventions: Device: PMMA IOL

INTERVENTIONS:
Device: Acrylic IOL — Acrylic IOL for long-term implantation in the cataract patient
  Other Names: AcrySof® Model MA30BA; AcrySof® Model MA60BM
  Arms: AcrySof IOL
Device: Silicone IOL — Silicone IOL for long-term implantation in the cataract patient
  Arms: Silicone IOL
Device: PMMA IOL — Polymethylmethacrylate IOL for long-term implantation in the cataract patient
  Arms: PMMA IOL

SUMMARY:
The purpose of this study is to compare the long-term visual acuity (VA) with an acrylic IOL to a silicone or polymethylmethacrylate (PMMA) IOL in cataract patients. This study will take place in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide voluntary consent and able to comprehend and sign the informed consent form;
* Pseudophakic patients implanted with an Acrylic (AcrySof®), PMMA or silicone IOL from 1994 to 2000;
* Clear intraocular media in study eye;
* Best-corrected visual acuity (decimal) within 3 months post-implantation of 0.8 (decimal VA chart) or more in study eye;
* No ocular or systemic condition which may affect visual acuity in study eye;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Complications that may impact visual acuity in study eye at the time of the prospective visit, such as glaucoma, diabetic retinitis, ocular inflammatory disease, retinal detachment, and others as specified in the protocol;
* Previous refractive surgery in study eye;
* Previous IOL exchange in study eye;
* Other protocol-specified exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Manager, Clinical Dev., Study Director — Alcon Japan, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11 study centers located in Japan.
Pre-assignment Details: Of the 104 enrolled, 6 subjects were exited as screen failures and deemed ineligible for participation. This reporting group includes all eligible subjects (98).
Groups:
- AcrySof: Acrylic IOL, prior implantation (1994-2000) in one or both eyes
- Silicone: Silicone IOL, prior implantation (1994-2000) in one or both eyes
- PMMA: Polymethylmethacrylate (PMMA) IOL, prior implantation (1994-2000) in one or both eyes
Period: Overall Study
Arm/Group | AcrySof | Silicone | PMMA
Started | 31 | 37 | 30
Completed | 31 | 37 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who used the study devices and underwent the long-term post-implantation visit examination (Safety Set).
Groups:
- PMMA: Polymethylmethacrylate IOL, prior implantation (1994-2000) in one or both eyes
- Total: Total of all reporting groups
Arm/Group | AcrySof | Silicone | PMMA | Total
Number analyzed (Participants) | 31 | 37 | 30 | 98
Age, Customized [Number; unit: subjects]
  <70 years | 2 | 4 | 6 | 12
  ≥70 and ≤79 years | 13 | 21 | 11 | 45
  ≥80 and ≤89 years | 12 | 12 | 9 | 33
  >90 years | 4 | 0 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 19 | 66
  Male | 8 | 13 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at the Long-Term, Post-Implantation Visit
Description: Measurement of best corrected (with spectacles or other visual corrective devices) visual acuity (at both near and distance). Visual Acuity (VA) is measured in logMAR (logarithm of the minimum angle of resolution). A lower logMAR value indicates better visual acuity. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (up to and including 3 months after implantation), long-term post-implantation visit (14-20 years after implantation)
Population: This analysis population includes all subjects who used the study devices and have data after implantation of study devices (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof | Silicone | PMMA
Number analyzed (Participants) | 31 | 37 | 30
logMAR
  Baseline | -0.06 (0.07) | -0.09 (0.07) | -0.07 (0.08)
  Change from baseline | 0.01 (0.08) | 0.04 (0.06) | -0.01 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study; retrospectively 14 to 20 years and prospectively for a single visit. This analysis group includes all subjects who used the study devices and underwent the long-term post-implantation visit examination. Ocular adverse events are presented for both study eye and non-study eye combined.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, whether or not related to the investigational medical device (test/control article or procedure). AEs are reported retrospectively (onset between Baseline (defined as the period within 3 months after surgery) and Informed Consent acquisition) and prospectively (onset after Informed Consent acquisition).
Groups:
- AcrySof (Retrospective): Subjects with prior implantation of acrylic IOL who experienced an AE related to decrease of BCVA in the study eye
- Silicone (Retrospective): Subjects with prior implantation of Silicone IOL who experienced an AE related to decrease of BCVA in the study eye
- PMMA (Retrospective): Subjects with prior implantation of PMMA IOL who experienced an AE related to decrease of BCVA in the study eye
- AcrySof (Prospective): Subjects with prior implantation of acrylic IOL who experienced an AE with onset after the Informed Consent acquisition
- Silicone (Prospective): Subjects with prior implantation of Silicone IOL who experienced an AE with onset after the Informed Consent acquisition
- PMMA (Prospective): Subjects with prior implantation of PMMA IOL who experienced an AE with onset after the Informed Consent acquisition
Arm/Group | AcrySof (Retrospective) | Silicone (Retrospective) | PMMA (Retrospective) | AcrySof (Prospective) | Silicone (Prospective) | PMMA (Prospective)
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/37 | 0/30 | 0/31 | 0/37 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 3/37 | 4/30 | 0/31 | 0/37 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AcrySof (Retrospective) (N=31) | Silicone (Retrospective) (N=37) | PMMA (Retrospective) (N=30) | AcrySof (Prospective) (N=31) | Silicone (Prospective) (N=37) | PMMA (Prospective) (N=30)
posterior capsule opacification (Eye disorders) | 0 | 3 | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.